CLINICAL TRIAL: NCT02372825
Title: Role of Free Iliac Crest Flap in Heel and Ankle Reconstruction
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Jussi Repo, Researcher, Helsinki University Central Hospital
Other Study IDs: 343/13/03/02/13/2
Record Dates: First submitted 2015-02-17; First posted 2015-02-26 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Limb Salvage
Keywords: Free iliac crest transfer; Bone reconstruction; Ankle reconstruction; Heel reconstruction
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Reconstructive surgery — Reconstructive surgery with the free iliac crest flap

SUMMARY:
Treatment of extensive traumatic acute bone defects or sequela in heel or ankle poses a formidable challenge for the reconstructive surgeon. These defects can be treated with the vascularized iliac crest transfer. The purpose of this study is to assess the reliability and the long-term outcomes of free iliac crest flap transfer for these indications.

DETAILED DESCRIPTION:
Thirteen patients were included in this study. Data was collected retrospectively from the patient records. The study design included three outcome measures to assess the clinical long-term outcomes. These were the Visual Analogue Scale Foot and Ankle (VAS FA), the Oswestry Disability Index (ODI), and the 15-dimensions (15D) health-related quality of life (HRQoL) instrument. The data was collected with postal approach and a written informed consent obtained from the seven participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute defects or sequela in the heel or ankle treated with the vascularized iliac crest transfer.

Exclusion Criteria:

1) Patients without treatment with the vascularized iliac crest transfer,

Exclusion criteria for the cross-sectional assessment:

1. deceased,
2. below-knee amputation,
3. permanent non-union

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirteen men patients with acute defects or sequela in the heel or ankle treated with the vascularized iliac crest transfer.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Heel and Ankle (VAS FA) | 2-26 years
  Assesses the function of the heel and ankle
Oswestry Disability Index (ODI) | 2-16 years
  Assesses the function of the donor site
The 15-Dimensions (15D) health-related quality of life (HRQoL) instrument | 2-26 years
  Assesses the HRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, MD, PhD, Study Director — Department of plastic and reconstructive surgery, HUCS
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland